CLINICAL TRIAL: NCT04230109
Title: A Phase 2 Study of Response-guided Neoadjuvant Sacituzumab Govitecan (IMMU-132) in Patients With Localized Triple-Negative Breast Cancer (NeoSTAR)
Brief Title: Sacituzumab Govitecan In TNBC
Acronym: NeoSTAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Laura M. Spring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-578
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Invasive Breast Cancer; Triple Negative Breast Cancer; ER-Negative Breast Cancer; PR-Negative Breast Cancer; HER2-negative Breast Cancer
Keywords: Invasive Breast Cancer; Triple Negative Breast Cancer; ER-Negative Breast Cancer; PR-Negative Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacituzumab Govitecan (monotherapy cohort) (Experimental): - The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Sacituzumab govitecan via iv, predetermined dosage per protocol, IV, 2 days per each 21-day cycle, for 4 cycles.
  * This can be followed by standard chemotherapy at the discretion of treating physician.
  Interventions: Drug: Sacituzumab Govitecan
- Sacituzumab Govitecan and Pembrolizumab (combination cohort) (Experimental): - The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Sacituzumab govitecan via iv, predetermined dosage per protocol, IV, 2 days per each 21-day cycle, for 4 cycles.
  * Pembrolizumab via iv, predetermined dosage per protocol, IV, 1 day per each 21-day cycle, for 4 cycles.
  * This can be followed by standard chemotherapy at the discretion of treating physician.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan via iv, predetermined dosage per protocol, two days per 21-day cycle, for 4 cycles (monotherapy cohort)
  Other Names: IMMU-132
Drug: Pembrolizumab — Pembrolizumab via iv, predetermined dosage per protocol, per 21-day cycle, for 4 cycles (combination cohort)
  Arms: Sacituzumab Govitecan and Pembrolizumab (combination cohort)

SUMMARY:
This research study is studying to evaluate sacituzumab govitecan for individuals with localized triple negative breast cancer (TNBC)

The names of the study drugs involved in this study is:

* Sacituzumab govitecan (SG)
* Pembrolizumab (combination therapy with SG)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

This research study involves an experimental study treatment. The names of the study drugs involved in this study is:

* Sacituzumab govitecan (SG)
* Pembrolizumab (combination therapy with SG)

The study is a umbrella study multi-arm phase II study of neoadjuvant SG-based therapy in patients with localized BC. The first cohort involves SG monotherapy. After the monotherapy cohort completes enrollment, the combination therapy cohort (SG with pembrolizumab) for patients with localized BC will open.

Future planned arms include SG with/without pembrolizumab for patients with Hormone Receptor positive (HR+) breast cancer and inflammatory breast cancer (IBC).

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* Eligible participants will receive Sacituzumab govitecan for up to 12 weeks.
* This can be followed by standard chemotherapy at the discretion of the treating physician.
* It is expected that about 50 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has not approved Sacituzumab govitecan as a treatment for patients with metastatic TNBC.

Sacituzumab govitecan (SG) is an antibody-drug conjugate which means it's made up of an antibody attached to an anticancer drug. An antibody is a protein normally made the immune system. Sacituzumab govitecan is believed to work by binding the antibody portion of the drug in the tumor(s) while the anticancer drug portion works to prevent cancer cells from growing/spreading.

After the SG monotherapy cohort completes enrollment, the combination therapy cohort (SG with immunotherapy) will open.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥ 18 years of age.
* Histologically confirmed diagnosis of invasive breast cancer, previously untreated.
* Participants must have biopsy proven ER negative (ER-), PR negative (PR-), HER2 negative (HER2-), invasive breast cancer. ER, PR, and HER2 positivity would be determined per ASCO/CAP guidelines by institutional (local) assessment. Patients with multi-focal and multicentric disease are eligible provided all histologically examined lesions are ER-/PR-/HER2- (local assessment). The need to biopsy additional lesions is at the discretion of the treating physician. Patients with bilateral invasive breast cancer are eligible provided all histologically examined lesions are ER-/PR-/HER2- (local assessment).
* Primary tumor (at least one lesion) 1 cm or greater measured by radiological imaging. Regional lymph node AJCC (v7) TNM stages N0-N2. If node positive, any primary tumor size is permissible. Absence of distant metastatic disease (AJCC TNM stage M0). Staging scans are not required and are per discretion of the treating physician.
* Pre- and postmenopausal women are eligible.
* ECOG performance status = 0, 1 (Karnofsky ≥60%, see Appendix A)
* Ability to understand and the willingness to sign a written informed consent form (ICF). Patient has signed the ICF prior to any screening procedures being performed and is able to comply with protocol requirements, including research biopsy.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:
* Absolute neutrophil count (ANC) ≥ 1,500 per mm3
* Platelets ≥ 100,000 per mm3
* Hemoglobin ≥9.0 g/dL
* INR ≤1.5
* Serum creatinine <1.5 mg/dL or creatinine clearance ≥50 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN.
* Total bilirubin ≤1.5 x ULN or in patients with well-documented Gilbert's Syndrome direct bilirubin ≤1.5 x ULN.

Exclusion Criteria:

* Inflammatory breast cancer, or locally recurrent breast cancer
* Participants currently receiving systemic therapy for any other malignancy or having received systemic therapy for a malignancy in the preceding 3 years.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia,or psychiatric illness/social situations that would limit compliance with study requirements.
* Clinically significant, uncontrolled heart disease and/or cardiac reppolarization abnormality including any of the following:

  * History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 6 months prior to study entry.
  * History of cardiac failure, known cardiomyopathy (LVEF < 50%; new LVEF assessment is not specifically required for this trial), significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:
* Known risk to prolong the QT interval or induce Torsade's de Pointes.
* Uncorrected hypomagnesemia or hypokalemia.
* Systolic Blood Pressure (SBP) >160 mmHg or <90 mmHg.
* Bradycardia (heart rate <50 at rest), by ECG or pulse. On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >470 screening ECG
* Pregnant or breast-feeding women are excluded from this study because the safety of study medications is not established.
* Known HIV-positive participants on combination antiretroviral therapy are ineligible.
* These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Separate HIV testing for this trial is not required. Similarly, separate Hepatitis B or C testing for this trial is not required, but patients with known (or history) of hepatitis B positive, or hepatitis C positive infection will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response(pCR) rate with sacituzumab govitecan | 12 Weeks
  pCR is defined as no residual invasive carcinoma in the breast and in the lymph node. The two-sided 95% CIs for pCR rate will be calculated.

SECONDARY OUTCOMES:
Disease-Free Survival | Time from the first dose of study treatment to disease recurrence/progression by RECIST v1.1 or death due to any cause, up to 36 months
  Kaplan-Meier methods and descriptive statistics
Overall Survival | defined as the time from the first dose of study treatment to the date of death or last contact up to 36 months
  Kaplan-Meier methods and descriptive statistics
Change in Breast Conserving Surgery Rate (BCS) rate | 12 Weeks
  RCB calculator: http:// RCB calculator: http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | Baseline to 12 weeks
  CTCAE v5.0
Assessment of Quality of life (QOL) | Baseline up to 12 Weeks
  EORTC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Laura Spring, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital - North Shore Cancer Center, Danvers, Massachusetts
  - Massachusetts General Hospital at Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Spring LM, Tolaney SM, Fell G, Bossuyt V, Abelman RO, Wu B, Maheswaran S, Trippa L, Comander A, Mulvey T, McLaughlin S, Ryan P, Ryan L, Abraham E, Rosenstock A, Garrido-Castro AC, Lynce F, Moy B, Isakoff SJ, Tung N, Mittendorf EA, Ellisen LW, Bardia A. Response-guided neoadjuvant sacituzumab govitecan for localized triple-negative breast cancer: results from the NeoSTAR trial. Ann Oncol. 2024 Mar;35(3):293-301. doi: 10.1016/j.annonc.2023.11.018. Epub 2023 Dec 12. PMID 38092228